CLINICAL TRIAL: NCT02491762
Title: The Effect of Breast Reconstruction Surgery Using Tissue Expanders on Respiratory Functions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yaron Har-Shai (Other)
Responsible Party: Sponsor-Investigator, Yaron Har-Shai, Clinical Professor Yaron Har-Shai, Carmel Medical Center
Organization: Carmel Medical Center (Other)
Other Study IDs: CMC-15-0029-CTIL
Record Dates: First submitted 2015-06-16; First posted 2015-07-08 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Function; Breast Reconstruction
Keywords: Serratus Anterior; Accessory Respiratory; Tissue Expander; Respiratory Function Tests
MeSH Terms: conditions — Respiratory Aspiration | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- bilateral: bilateral breast construction candidates will go through respiratory function tests a month prior to surgery, a month after surgery and three months after surgery
  Interventions: Procedure: respiratory function tests
- unilateral: unilateral breast construction candidates will go through respiratory function tests a month prior to surgery, a month after surgery and three months after surgery
  Interventions: Procedure: respiratory function tests

INTERVENTIONS:
Procedure: respiratory function tests — FVC, FEV1, MVV, FRC, RV, TLC, MIP, MEP

SUMMARY:
This study evaluates the effect of breast reconstruction surgery on respiratory functions. 45 patients elected for unilateral or bilateral breast reconstruction surgery will go through respiratory function examinations a month prior to the surgery, one month after surgery and three months after surgery.

DETAILED DESCRIPTION:
Breast reconstruction surgery using tissue expander and implant technique is the most common breast reconstruction surgery. During this procedure, the surgeon will insert a silicone expander under the Pectoralis Major muscle. In order to fully cover the expander, the surgeon will detach the Serratus Anterior [SA] muscle from its natural attachments in the rib cage and will attach the free edges to the lateral edge of the Pectoralis Major muscle. After the wound is healed, a gradual inflation of the expander with a physiological fluid will be done by injecting the fluid into a subcutaneous filling port connected to the expander by silicone tubing. When the tissues around the expander will reach the required size, the tissue expander can be replaced by a permanent silicone implant.

The SA attachments are to the superior angle, medial border and inferior angle of the scapula and to the first to eighth ribs. Its main functions are stabilization and protraction of the scapula and turning the glenoid cavity superiorly in abduction of arms. In addition, the SA is an accessory respiratory muscle: when the scapula is stabilized, its contraction will lift the rib cage in order to help breathing. The importance of the SA in breathing has been examined since the late 19th century and until this day it is not fully agreed upon. Most studies agree that the SA major role in breathing is in deep breaths and is that the muscle is most effective for this purpose when arms are lifted.

Since breast reconstruction procedure includes detachment of the SA from the rib cage and there by canceling its respiratory function, an examination of the respiratory functions before and after the procedure is in order to determine whether or not the overall respiratory functions had been effected.

45 patients elected for unilateral or bilateral breast reconstruction surgery will go through respiratory function examinations a month prior to the surgery, one month after surgery and three months after surgery. The examinations will include the following tests: Spirometry: FVC, FEV1, MVV. Lung capacities: FRC, RV, TLC. Breathing muscle strength: MIP, MEP.

ELIGIBILITY:
Inclusion Criteria:

* all subjects were elected for a unilateral or bilateral breast reconstruction using tissue expander by the Oncoplastic Committee of the plastic surgery unit in Carmel Medical Center.
* all subjects agrees to enroll in research

Exclusion Criteria:

* subject is in a mental or physical condition that does not allow her to go through respiratory function tests.
* subject was found with a respiratory disfunction or disease in the first respiratory function tests.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients elected for breast reconstruction surgery using tissue expander-implant technique
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity -FVC | a month prior to surgery
  Forced vital capacity: the determination of the vital capacity from a maximally forced expiratory effort
Forced expiratory volume at one second -FEV1 | a month prior to surgery
  Volume that has been exhaled at the end of the first second of forced expiration
Maximum voluntary ventilation-MVV | a month prior to surgery
  Maximal voluntary ventilation: volume of air expired in a specified period during repetitive maximal effort
Functional residual capacity-FRC | a month prior to surgery
  Functional residual capacity: the volume in the lungs at the end-expiratory position
Residual volume -RV | a month prior to surgery.
  Residual volume: the volume of air remaining in the lungs after a maximal exhalation.
Total lung capacity-TLC | a month prior to surgery.
  Total lung capacity: the volume in the lungs at maximal inflation, the sum of VC and RV.
Maximal inspiratory pressure-MIP | a month prior to surgery.
  Maximal inspiratory pressure (MIP) is the maximal pressure that can be produced by the patient trying to inhale through a blocked mouthpiece
Maximal expiratory pressure-MEP | a month prior to surgery.
  Maximal expiratory pressure (MEP) is the maximal pressure measured during forced expiration (with cheeks bulging) through a blocked mouthpiece after a full inhalation.
Forced vital capacity -FVC | a month after surgery
  Forced vital capacity: the determination of the vital capacity from a maximally forced
Forced vital capacity -FVC | three months after surgery
  Forced vital capacity: the determination of the vital capacity from a maximally forced
Forced expiratory volume at one second -FEV1 | a month after surgery
  Volume that has been exhaled at the end of the first second of forced expiration
Forced expiratory volume at one second -FEV1 | three months after surgery
  Volume that has been exhaled at the end of the first second of forced expiration
Maximum voluntary ventilation-MVV | a month after surgery
  Maximal voluntary ventilation: volume of air expired in a specified period during repetitive maximal effort
Maximum voluntary ventilation-MVV | three months after surgery
  Maximal voluntary ventilation: volume of air expired in a specified period during repetitive maximal effort
Functional residual capacity-FRC | a month after surgery
  Functional residual capacity: the volume in the lungs at the end-expiratory position
Functional residual capacity-FRC | three months after surgery
  Functional residual capacity: the volume in the lungs at the end-expiratory position
Residual volume -RV | a month after surgery
  Residual volume: the volume of air remaining in the lungs after a maximal exhalation.
Residual volume -RV | three months after surgery
  Residual volume: the volume of air remaining in the lungs after a maximal exhalation.
Total lung capacity-TLC | a month after surgery.
  Total lung capacity: the volume in the lungs at maximal inflation, the sum of VC and RV.
Total lung capacity-TLC | three months after surgery.
  Total lung capacity: the volume in the lungs at maximal inflation, the sum of VC and RV.
Maximal inspiratory pressure-MIP | a month after surgery
  Maximal inspiratory pressure (MIP) is the maximal pressure that can be produced by the patient trying to inhale through a blocked mouthpiece
Maximal inspiratory pressure-MIP | three months after surgery.
  Maximal inspiratory pressure (MIP) is the maximal pressure that can be produced by the patient trying to inhale through a blocked mouthpiece
Maximal expiratory pressure-MEP | a month after surgery.
  Maximal expiratory pressure (MEP) is the maximal pressure measured during forced expiration (with cheeks bulging) through a blocked mouthpiece after a full inhalation.
Maximal expiratory pressure-MEP | three months after surgery.
  Maximal expiratory pressure (MEP) is the maximal pressure measured during forced expiration (with cheeks bulging) through a blocked mouthpiece after a full inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Har-Shai, Proffesor, Principal Investigator — Carmel Medical Center-Israel
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Terakado S, Takeuchi T, Miura T, Sato H, Nishioka N, Fujieda Y, Kobayashi R, Ibukiyama C. Early occurrence of respiratory muscle deoxygenation assessed by near-infrared spectroscopy during leg exercise in patients with chronic heart failure. Jpn Circ J. 1999 Feb;63(2):97-103. doi: 10.1253/jcj.63.97. PMID 10084371
- [Background] Legrand R, Marles A, Prieur F, Lazzari S, Blondel N, Mucci P. Related trends in locomotor and respiratory muscle oxygenation during exercise. Med Sci Sports Exerc. 2007 Jan;39(1):91-100. doi: 10.1249/01.mss.0000241638.90348.67. PMID 17218889
- [Background] Legrand R, Prieur F, Marles A, Nourry C, Lazzari S, Blondel N, Mucci P. Respiratory muscle oxygenation kinetics: relationships with breathing pattern during exercise. Int J Sports Med. 2007 Feb;28(2):91-9. doi: 10.1055/s-2006-924056. Epub 2006 Jul 12. PMID 16838222
- [Background] Lomax M, Tasker L, Bostanci O. An electromyographic evaluation of dual role breathing and upper body muscles in response to front crawl swimming. Scand J Med Sci Sports. 2015 Oct;25(5):e472-8. doi: 10.1111/sms.12354. Epub 2014 Dec 30. PMID 25640018
- [Background] Machado de Sousa O, Costacurta L. Electromyographic study of the M. serratus anterior during respiration. Electromyogr Clin Neurophysiol. 1984 Nov-Dec;24(7):547-59. No abstract available. PMID 6510353
- [Background] Mancini DM, Ferraro N, Nazzaro D, Chance B, Wilson JR. Respiratory muscle deoxygenation during exercise in patients with heart failure demonstrated with near-infrared spectroscopy. J Am Coll Cardiol. 1991 Aug;18(2):492-8. doi: 10.1016/0735-1097(91)90605-9. PMID 1856417
- [Background] Matusiewicz AK, Carter AE, Landes RD, Yi R. Statistical equivalence and test-retest reliability of delay and probability discounting using real and hypothetical rewards. Behav Processes. 2013 Nov;100:116-22. doi: 10.1016/j.beproc.2013.07.019. Epub 2013 Aug 14. PMID 23954833
- [Background] Moalla W, Dupont G, Berthoin S, Ahmaidi S. Respiratory muscle deoxygenation and ventilatory threshold assessments using near infrared spectroscopy in children. Int J Sports Med. 2005 Sep;26(7):576-82. doi: 10.1055/s-2004-830332. PMID 16195992
- [Background] Ogata H, Arimitsu T, Matsuura R, Yunoki T, Horiuchi M, Yano T. Relationship between oxygenation in inactive biceps brachii muscle and hyperventilation during leg cycling. Physiol Res. 2007;56(1):57-65. doi: 10.33549/physiolres.930888. Epub 2006 Feb 23. PMID 16497096
- [Background] Ogata H, Reyihan A, Yano T. Kinetics of oxygenation in inactive forearm muscle during ramp leg cycling. J Physiol Anthropol Appl Human Sci. 2004 Jan;23(1):7-17. doi: 10.2114/jpa.23.7. PMID 14757996
- [Background] Reid DC, Bowden J, Lynne-Davies P. Role of selected muscles of respiration as influenced by posture and tidal volume. Chest. 1976 Nov;70(5):636-40. doi: 10.1378/chest.70.5.636. PMID 975981
- [Background] TOKIZANE T, KAWAMATA K, TOKIZANE H. Electromyographic studies on the human respiratory muscles; studies on the activity pattern of neuromuscular units. Jpn J Physiol. 1952 Feb;2(3):232-47. doi: 10.2170/jjphysiol.2.232. No abstract available. PMID 14927261
- [Background] Tsoi B, Ziolkowski NI, Thoma A, Campbell K, O'Reilly D, Goeree R. Systematic review on the patient-reported outcomes of tissue-expander/implant vs autologous abdominal tissue breast reconstruction in postmastectomy breast cancer patients. J Am Coll Surg. 2014 May;218(5):1038-48. doi: 10.1016/j.jamcollsurg.2014.02.011. Epub 2014 Feb 19. No abstract available. PMID 24745568
- [Background] Wang L, Yoshikawa T, Hara T, Nakao H, Suzuki T, Fujimoto S. Which common NIRS variable reflects muscle estimated lactate threshold most closely? Appl Physiol Nutr Metab. 2006 Oct;31(5):612-20. doi: 10.1139/h06-069. PMID 17111016
- [Background] Cannon DT, Grout SL, May CA, Strom SD, Wyckoff KG, Cipriani DJ, Buono MJ. Recruitment of the serratus anterior as an accessory muscle of ventilation during graded exercise. J Physiol Sci. 2007 Apr;57(2):127-31. doi: 10.2170/physiolsci.RP001807. Epub 2007 Apr 6. PMID 17408533
- [Background] Cerqueira EP, Garbellini D. Electromyographic study of the pectoralis major, serratus anterior and external oblique muscles during respiratory activity in humans. Electromyogr Clin Neurophysiol. 1999 Apr-May;39(3):131-7. PMID 10228878
- [Background] Chawla AK, Kachnic LA, Taghian AG, Niemierko A, Zapton DT, Powell SN. Radiotherapy and breast reconstruction: complications and cosmesis with TRAM versus tissue expander/implant. Int J Radiat Oncol Biol Phys. 2002 Oct 1;54(2):520-6. doi: 10.1016/s0360-3016(02)02951-6. PMID 12243831
- [Background] Fischer JP, Wes AM, Nelson JA, Basta M, Rohrbach JI, Wu LC, Serletti JM, Kovach SJ. Propensity-matched, longitudinal outcomes analysis of complications and cost: comparing abdominal free flaps and implant-based breast reconstruction. J Am Coll Surg. 2014 Aug;219(2):303-12. doi: 10.1016/j.jamcollsurg.2014.02.028. Epub 2014 Apr 8. PMID 24916480
- [Background] Gallistel CR. The importance of proving the null. Psychol Rev. 2009 Apr;116(2):439-53. doi: 10.1037/a0015251. PMID 19348549
- [Background] GRONBAEK P, SKOUBY AP. The activity pattern of the diaphragm and some muscles of the neck and trunk in chronic asthmatics and normal controls. A comparative electromyographic study. Acta Med Scand. 1960 Dec 20;168:413-25. doi: 10.1111/j.0954-6820.1960.tb06672.x. No abstract available. PMID 13708898
- [Background] JEFFERSON NC, OGAWA T, SYLEOS C, ZAMBETOGLOU A, NECHELES H. Restoration of respiration by nerve anastomosis. Am J Physiol. 1960 May;198:931-3. doi: 10.1152/ajplegacy.1960.198.5.931. No abstract available. PMID 14407006
- [Background] Johnson BD, Babcock MA, Suman OE, Dempsey JA. Exercise-induced diaphragmatic fatigue in healthy humans. J Physiol. 1993 Jan;460:385-405. doi: 10.1113/jphysiol.1993.sp019477. PMID 8487201